CLINICAL TRIAL: NCT04945824
Title: An Open-label, Multi-center, Bilateral, Human Factors Study to Evaluate the Utilization and Safety of a Novel Intracanalicular Insertion Device in Healthy Subjects
Brief Title: A Human Factors Study to Evaluate a Novel Intracanalicular Insertion Device in Healthy Subjects
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: inserter device did not perform as expected
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OTX-DPI-2020-401
Record Dates: First submitted 2021-06-01; First posted 2021-06-30 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Novel Intracanalicular Insertion Device (Experimental)
  Interventions: Drug: Dexamethasone Ophthalmic; Device: Dilator

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic — Insertion Device: A handheld mechanical device used by the clinician to dilate the punctum and deliver the DEXTENZA insert into the canaliculus; designed to be single-use and pre-loaded with a single DEXTENZA insert.
Device: Dilator — Intracanalicular Dilator Device

SUMMARY:
This is an open-label, multi-center, bilateral, human factors study designed to evaluate the utilization and safety of a novel intracanalicular insertion device in healthy subjects and to evaluate the concentration of DEXTENZA in tears. Each subject's participation is expected to last for approximately 1 month from the DEXTENZA insertion.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy adult subject aged 18 years or older with no known significant health problems
* Are willing to refrain from wearing contact lens for the duration of the study
* Are willing and able to comply with clinic visits and study related procedures
* Are willing and able to sign the informed consent form

Exclusion Criteria:

* Have known significant health problems
* Are women of reproductive potential
* Are breastfeeding
* Are a known steroid responder
* Have a history of herpes simplex virus keratitis or present active bacterial, viral, or fungal keratitis in either eye
* Have a history of complete punctal occlusion in one or both punctum
* Currently use topical ophthalmic steroid medications
* Are unwilling or unable to comply with the study protocol
* Are determined by the Investigator to not be included for reasons not already specified (e.g., systemic, behavioral, or other ocular

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Ease of insertion as assessed by Post-Insertion Investigator Questionnaire | Assessed at Visit 1 (Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Ocular Therapeutix, Inc., Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided